CLINICAL TRIAL: NCT01274598
Title: Open Label Study to Evaluate the Safety of Lactobacillus Rhamnosus GG ATCC 53103 (LGG) in Elderly Subjects
Brief Title: Study to Evaluate the Safety of Lactobacillus Rhamnosus GG ATCC 53103 (LGG) in Elderly Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Patricia L. Hibberd, Chief, Division of Global Health; Department of Pediatrics, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: U01AT002952-01A2 (NIH)
Record Dates: First submitted 2011-01-03; First posted 2011-01-11 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2017-01

CONDITIONS: Healthy; Elderly
Keywords: Probiotics; Safety; Elderly; Lactobacillus; LGG

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lactobacillus Rhamnosus GG, ATCC 53103 (LGG) (Experimental): Lactobacillus rhamnosus GG ATCC 53103 1 x 10^10 twice a day for 28 days
  Interventions: Biological: Lactobacillus Rhamnosus GG, ATCC 53103 (LGG)

INTERVENTIONS:
Biological: Lactobacillus Rhamnosus GG, ATCC 53103 (LGG) — 1x10^10 CFU by mouth twice daily for 28 days
  Other Names: Culturelle

SUMMARY:
This is a phase I, open label clinical trial to evaluate the safety of Lactobacillus rhamnosus GG (LGG) in elderly subjects. Lactobacilli are part of the normal flora of the intestine. LGG is one of several strains of Lactobacilli that is used as a probiotic or microorganism administered to confer "health benefits". Our research is focused on studying the possible therapeutic effects of LGG. The study hypotheses are:

* LGG administered twice daily will be safe and well tolerated in elderly subjects
* LGG will colonize the stool of elderly subjects and will modify the diversity and richness of the microbiota in their nasopharyngeal and stool specimens

ELIGIBILITY:
Inclusion Criteria:

1. Age 65-80 years
2. Willing to complete the informed consent process
3. Able and willing to participate for the planned duration of the study, including availability for follow-up telephone contact
4. Willing to comply with protocol and report on compliance and side effects during the study period
5. Informed consent obtained and signed prior to screening

Exclusion Criteria:

1. Consumption of supplements or food products containing LGG or probiotics for 28 days prior to the start of the study or consumption of yogurt that has the "live and active cultures" seal.
2. Known or suspected allergies to probiotics, Lactobacillus, microcrystalline cellulose, gelatin, or antibiotics that may be used to treat LGG bacteremia or infection (i.e., subject able to tolerate at least 2 of the following regimens - Ampicillin or other beta lactam antibiotic, and Clindamycin, and Moxifloxacin).
3. Received oral or parenteral antibiotics within 4 weeks of enrollment or prescribed antibiotics on the day of enrollment
4. Drug or alcohol abuse within the previous 12 months
5. Hospitalization, major surgery or endoscopy within the last 3 months
6. Scheduled hospital admission within 3 months of enrollment
7. Resident of a nursing home or rehabilitation center
8. Presence of any of the following:

   * Grade 2 or higher abnormal vital signs or abnormalities on physical exam
   * Indwelling catheter or implanted hardware/prosthetic device or feeding tube
   * Active bowel leak, acute abdomen, colitis, or active GI disease or history of gastric or intestinal dysmotility, slowed transit time, variable small intestinal permeability, pancreatitis, history of gastrointestinal tract cancer or inflammatory bowel disease
   * History of Hepatitis B or Hepatitis C infections, cirrhosis, or chronic liver disease
   * Underlying structural heart disease such as abnormal native heart valve or congenital abnormality, previous history of endocarditis or valve replacement, Stage IV congestive heart failure
   * History of peripheral vascular disease or stroke
   * Immunosuppression including HIV positive, solid organ or stem cell transplant recipient, receiving any oral or parenteral immunosuppressive therapy, neutrophil count <500/mm3, or an anticipated drop in the neutrophil count to <500/mm3 or active or planned chemotherapy or radiotherapy
   * History of collagen vascular or autoimmune disease
   * End stage renal disease
   * History of chronic obstructive pulmonary disease or asthma
   * Diabetes or thyroid disease
   * Active TB
9. Positive drug or alcohol testing at screening or positive breathalyzer at baseline or an unwillingness to undergo drug and alcohol testing
10. Abnormal laboratory tests defined as any of the following:

    * White blood cell (WBC) < 3.3 or > 12.0 K/µL
    * Platelets < 125 K/µL
    * Hemoglobin Males: < 12.0 g/dL; Females: < 11.0 g/dL
    * Creatinine > 1.8 mg/dL
    * Blood urea nitrogen (BUN) >27 mg/dL
    * Aspartate aminotransferase (AST) > 1.25 ULN
    * Alanine aminotransferase (ALT) > 1.25 ULN
    * Alkaline phosphatase > 2.0 ULN
    * Bilirubin (total) > 1.5 ULN
    * Glucose (non-fasting ) >126 mg/dL
    * Positive HIV, Hepatitis B surface antigen or Hepatitis C antibody
11. Any other condition that in the opinion of the investigator would jeopardize the safety or rights of the subject participating in the study or would make it unlikely the subject could complete the study

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 15 (Actual)
Dates: Start 2010-12; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Occurrence of adverse events that are possibly or probably related to administration of LGG | through day 56
  Adverse events will be detected during study visits with standardized questionnaires, medical history, vital signs, physical examinations, laboratory tests and review of subject diaries as well as between study visits on telephone calls based on responses to adverse event questionnaires.

SECONDARY OUTCOMES:
Changes in the richness and bacterial diversity of the nasopharyngeal and gut microbiota and presence of LGG in stool specimens by routine culture | through day 56
  We will analyze the stool and nasopharyngeal samples to learn what bacteria are present during different phases of the study and how the types and quantities of bacteria may change over time.

CONTACTS AND LOCATIONS:
Overall Officials: Patricia L Hibberd, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Solano-Aguilar G, Molokin A, Botelho C, Fiorino AM, Vinyard B, Li R, Chen C, Urban J Jr, Dawson H, Andreyeva I, Haverkamp M, Hibberd PL. Transcriptomic Profile of Whole Blood Cells from Elderly Subjects Fed Probiotic Bacteria Lactobacillus rhamnosus GG ATCC 53103 (LGG) in a Phase I Open Label Study. PLoS One. 2016 Feb 9;11(2):e0147426. doi: 10.1371/journal.pone.0147426. eCollection 2016. PMID 26859761
- [Derived] Hibberd PL, Kleimola L, Fiorino AM, Botelho C, Haverkamp M, Andreyeva I, Poutsiaka D, Fraser C, Solano-Aguilar G, Snydman DR. No evidence of harms of probiotic Lactobacillus rhamnosus GG ATCC 53103 in healthy elderly-a phase I open label study to assess safety, tolerability and cytokine responses. PLoS One. 2014 Dec 1;9(12):e113456. doi: 10.1371/journal.pone.0113456. eCollection 2014. PMID 25438151